CLINICAL TRIAL: NCT04292496
Title: Efifcacy and Safety of Anastomotic Leak Testing in Gastric Cancer: a Randomized Controlled Trial
Brief Title: Anastomotic Leak Testing in Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Yunhong Tian, Professor, Nanchong Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020001
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Anastomotic Leak; Gastric Cancer; Surgery; Testing, Reality; Gastroscopy
Keywords: Anastomotic leakage; Gastric cancer; Leakage testing; Total gastrectomy; Gastroscopy
MeSH Terms: conditions — Anastomotic Leak; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraperative leak testing group (Experimental): i) the integrity of the anastomosis can be directly observed under gastroscopy. ii) the distal of Roux limb was temporarily blocked, then the bowel of anastomosis was inflated by air, following 60 milliliter methylene blue.
  Interventions: Procedure: Introperative leak testing
- Non-intraoperative leak testing group (No Intervention): Non intraoperative leak testing was performed intraoperatively.

INTERVENTIONS:
Procedure: Introperative leak testing — After anastomosis was completed. We test the integrity of anastomosis intraoperatively.
  Arms: Intraperative leak testing group

SUMMARY:
Anastomotic leak after radical gastrectomy is a serious complication. Intraoperative leak testing was often used to assess the integrity of the anastomosis. However, the reliability, clinical benefits and safety of intraoperative leak testing are controversial. Our aim is to evaluate the effect and safety of intraoperative leak testing, and to compare the surgical complications of patients in intraoperative leak testing group with patients in non-intraoperative leak testing group.

DETAILED DESCRIPTION:
Anastomotic leak after radical gastrectomy is a serious complication. Intraoperative leak testing was often used to assess the integrity of the anastomosis. However, the reliability, clinical benefits and safety of intraoperative leak testing are controversial. Our aim is to evaluate the effect and safety of intraoperative leak testing, and to compare the surgical complications of patients in intraoperative leak testing group with patients in non-intraoperative leak testing group. patients underwent total gastrectomy for gastric cancer, with esophagojejunostomy reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. resectable gastric carcinoma according to the eighth edition of the TNM (clinical stages I-III).
2. Eastern Cooperative Oncology Group performance status of 0 or 1.
3. American Society of Anesthesiologists class of I-III.

Exclusion Criteria:

1. Patients had distant metastasis.
2. presence of obvious contraindications to surgery (e.g., liver and/or kidney function abnormalities).
3. any participation in another clinical trial within the past 6 months.
4. Previous chemotherapy or radiation therapy for any other malignancies.
5. past history of gastric resection, gastric cancer-related complications, other malignancy diagnosed within the previous 5 years,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage | 2 months
  all patients underwent upper gastrointestinal radiography after surgery for detecting the integrity of anastomosis. X-ray to detect the integrity of the anastomosis

SECONDARY OUTCOMES:
Postoperative surgical complications | 3 months
  Any surgical complication that occured postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China

REFERENCES:
- [Derived] Gao Z, Luo H, Ma L, Bai D, Qin X, Bautista M, Gong L, Peng Y, Hu J, Tian Y. Efficacy and safety of anastomotic leak testing in gastric cancer: a randomized controlled trial. Surg Endosc. 2023 Jul;37(7):5265-5273. doi: 10.1007/s00464-023-10025-w. Epub 2023 Mar 27. PMID 36971816
- Available data/document: Study Protocol — https://doi.org/10.1007/s00464-023-10025-w